CLINICAL TRIAL: NCT05648669
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of Elagolix in Patients With Moderate to Severe Endometriosis-Associated Pain
Brief Title: A Study to Evaluate Safety and Efficacy of Elagolix in Patients With Moderate to Severe Endometriosis-Associated Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL-YH001-002
Record Dates: First submitted 2022-11-16; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elagolix (Experimental): Elagolix 200 mg twice daily (BID) for the 6-month Treatment Period
  Interventions: Drug: Elagolix
- Elagolix placebo (Placebo Comparator): Placebo BID for the 6-month Treatment Period
  Interventions: Drug: Elagolix placebo

INTERVENTIONS:
Drug: Elagolix — 200 mg tablet
  Arms: Elagolix
Drug: Elagolix placebo — Elagolix-matched Placebo tablet
  Arms: Elagolix placebo

SUMMARY:
This is a Phase 3, multicenter, double-blind, placebo-controlled, randomized study to assess the safety and efficacy of elagolix versus placebo in premenopausal 18 to 49 year old women with moderate to severe endometriosis-associated pain.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, double-blind, placebo-controlled, randomized study to assess the safety and efficacy of elagolix versus placebo in premenopausal 18 to 49 year old women with moderate to severe endometriosis-associated pain. Participants will be randomised in a 1:1 ratio to receive either elagolix ( 200mg )or placebo. Participants will be administered the study drug up to month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Participant understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent.
2. Participant is premenopausal female, between 18 and 49 years of age (both inclusive), regular menstruation within 3 months before screening.
3. Participant clinical diagnosis of endometriosis (laparoscopy or laparotomy) performed within 10 years of entry into Screening.
4. Participant agrees to use non-hormonal contraception from signing the informed consent through 30 days after last dose of investigational product.
5. Participant cervical smear is normal or abnormal without clinical significance (normal cervical smear within 6 months prior to screening; or participant is virgin and decides not to undergo cervical smear); Atypical Squamous Cells of Undetermined Significance (ASCUS) may be combined with human papillomavirus (HPV) testing. ASCUS participants may be included if they are negative for high-risk HPV.
6. Participant who is 40 years or older in age has a normal or abnormal without clinical significance mammogram at screening or within 6 months prior to screening [Breast Imaging Reporting Data System (BI-RADS) classification 1-3 or equivalent].

Exclusion Criteria:

1. Participant who has a history of sensitivity to elagolix or excipients.
2. Participant who blood pregnancy test is positive at screening or on the day of randomization.
3. Participant who has an intra-uterine device (IUD) or contraceptive sub-dermal implant (If the IUD or sub-dermal implant is removed at least 30 days, participant may be screened for the study).
4. Participant who has a history of drug or alcohol abuse within 6 months of screening.
5. Participant who is hepatitis B patient [hepatitis B surface antigen (HbsAg) positive and detection of HBV-DNA suggests viral replication]; hepatitis C patients [hepatitis C virus (HCV) antibody positive and detection of HCV-RNA suggests viral replication]; syphilis screening positive (except for specific antibody detection positive, non-specific antibody detection negative and confirmed as inactive infection in combination with clinical judgment), known history of human immunodeficiency virus (HIV) positive or HIV screening positive;
6. Participant who has used moderate or strong inducers of cytochrome P450 3A or inhibitors of organic anion transporting polypeptide 1B1 (OATP1B1) within 30 days prior to first dose.
7. Participant who has unstable medical diseases in the opinion of the investigator (e.g. uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled seizures, angina unstable, inflammatory bowel disease, hyperprolactinemia, malignancy, or significant infection).
8. Participant who has a history of major depression or post-traumatic stress disorder within 2 years of screening or a history of other major psychiatric disorder.
9. Participant who has a history of surgical history of hysterectomy, bilateral oophorectomy, procedure that interferes with gastrointestinal mo
10. Participant who in the opinion of the investigator has a history of previous non-response to gonadotropin-releasing hormone agonists, antagonists. tility, any recent major or minor surgery.
11. Participant who need to use rescue analgesic drugs other than those specified in the protocol, or disagree to use rescue analgesic drugs specified in the protocol during the screening period and treatment period.
12. Participant who has any other chronic pain syndrome that requires chronic analgesic or other chronic therapy, which, in the opinion of the investigator, would interfere with the assessment of endometriosis-related pain.
13. Participant who has used of any systemic steroids for more than 2 weeks within 3 months prior to screening or is likely to require such treatment during the course of the study. Over-the-counter and prescription topical, inhaled or nasal corticosteroids are allowed.
14. Participant who has participated in another investigational study or treatment within 30 days prior to first dose.
15. Participant who has previously participated in an elagolix study.
16. Participant who has a of abnormal uterine or vaginal bleeding within 3 months prior to Screening.
17. Participant who has a history or presence of osteoporosis or other metabolic bone, or clinically significant hypocalcemia, hypo- or hyperphosphatemia at screening.
18. Participant who has dual-energy x-ray (DXA) absorptiometry scan results of the lumbar spine (L1-L4), femoral neck, or total hip bone mineral density (BMD) below normal 2.0 or more at screening (Z-score for patients < 40 years, T-score for patients ≥ 40 years).
19. Participant who may increase study-related risks or interfere with the interpretation of study results in the opinion of the investigator, who are considered unsuitable for enrollment by the investigator and/or the sponsor.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Estimated)
Dates: Start 2022-09-04 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders of Dysmenorrhea (DYS) at week 12 | Week12
  The criteria for a responder was based on a pre-defined threshold.
Percentage of Responders of Non-Menstrual Pelvic Pain (NMPP) at week 12 | Week12
  The criteria for a responder was based on a pre-defined threshold.

SECONDARY OUTCOMES:
Safety Specifications in the Treatment Period | Baseline, Week24
  Adverse event and serious adverse event
Change in Numeric Rating Scale (NRS) Scores at week 12 | Week12
  The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Change in Dysmenorrhea (DYS) Score at week 24 | Week24
  The DYS pain scale ranges from none to severe.
Change in Non-Menstrual Pelvic Pain (NMPP) Score at week 24 | Week24
  The NMPP pain scale ranges from none to severe.

CONTACTS AND LOCATIONS:
Overall Officials: jinhua Leng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China